CLINICAL TRIAL: NCT02343614
Title: Celecoxib for the Treatment of Non-muscle Invasive Bladder Cancer
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Azienda Ospedaliero-Universitaria Consorziale Policlinico di Bari (Other)
Responsible Party: Principal Investigator, Pagliarulo Vincenzo, Medical Doctor, Azienda Ospedaliero-Universitaria Consorziale Policlinico di Bari
Allocation: Not Applicable | Model: Single Group | Masking: Single | Purpose: Treatment
Other Study IDs: 2401
Record Dates: First submitted 2015-01-16; First posted 2015-01-22 (Estimated); Last update posted 2015-01-22 (Estimated); Status verified 2015-01

CONDITIONS: Non Muscle Invasive Bladder Cancer
Keywords: Intermediate risk; Cox-2 inhibitors
MeSH Terms: conditions — Non-Muscle Invasive Bladder Neoplasms | interventions — Celecoxib

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- ARM A (Experimental): Patients undergoing treatment with oral celecoxib
  Interventions: Drug: Celecoxib

INTERVENTIONS:
Drug: Celecoxib

SUMMARY:
The treatment of non-muscle invasive bladder cancer (NMIBC) is problematic given the variable natural history of the disease. Although contemporary treatment options are limited, new targets and new approaches are under investigation for preventing bladder cancer recurrence and progression. Among those, COX-2 is a promising target since plays an important role in urothelial carcinogenesis and iCOX-2 selective inhibitors, like celecoxib, effectively inhibit tumor development and growth and enhances survival, in bladder cancer in vitro and in vivo models.

Therefore, the investigators conducted a pilot study of celecoxib to prevent recurrence in patients with intermediate risk NMIBC.

ELIGIBILITY:
Inclusion Criteria:

* Histologically proven urothelial bladder cancer
* Intermediate risk NMIBC
* ECOG Performance Status ≤ 2 or Karnofsky Score ≥ 60%
* Imaging study excluding upper urinary tract TCC

Exclusion Criteria:

* Pregnant and lactating women;
* Advanced co-existing medical or psychiatric disorders;
* Positive history of gastro-intestinal disease (peptic ulcer, inflammatory disease), intestinal bleeding;
* History of allergy to sulfonamide drugs;
* Concomitant investigational medications.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 58 (Actual)
Dates: Start 2003-03; Primary Completion 2013-10 (Actual); Study Completion 2014-01 (Actual)

PRIMARY OUTCOMES:
Time to first recurrence | 5 years
Safety assessed by description of grade 1-4 adverse events | 5 years

CONTACTS AND LOCATIONS:
Overall Officials: Vincenzo VP Pagliarulo, Medical Doctor, Principal Investigator — Azienda Ospedaliero-Universitaria Consorziale Policlinico di Bari

REFERENCES:
- [Background] Arber N, Eagle CJ, Spicak J, Racz I, Dite P, Hajer J, Zavoral M, Lechuga MJ, Gerletti P, Tang J, Rosenstein RB, Macdonald K, Bhadra P, Fowler R, Wittes J, Zauber AG, Solomon SD, Levin B; PreSAP Trial Investigators. Celecoxib for the prevention of colorectal adenomatous polyps. N Engl J Med. 2006 Aug 31;355(9):885-95. doi: 10.1056/NEJMoa061652. PMID 16943401
- [Background] Bertagnolli MM, Eagle CJ, Zauber AG, Redston M, Solomon SD, Kim K, Tang J, Rosenstein RB, Wittes J, Corle D, Hess TM, Woloj GM, Boisserie F, Anderson WF, Viner JL, Bagheri D, Burn J, Chung DC, Dewar T, Foley TR, Hoffman N, Macrae F, Pruitt RE, Saltzman JR, Salzberg B, Sylwestrowicz T, Gordon GB, Hawk ET; APC Study Investigators. Celecoxib for the prevention of sporadic colorectal adenomas. N Engl J Med. 2006 Aug 31;355(9):873-84. doi: 10.1056/NEJMoa061355. PMID 16943400
- [Background] Bombardier C, Laine L, Reicin A, Shapiro D, Burgos-Vargas R, Davis B, Day R, Ferraz MB, Hawkey CJ, Hochberg MC, Kvien TK, Schnitzer TJ; VIGOR Study Group. Comparison of upper gastrointestinal toxicity of rofecoxib and naproxen in patients with rheumatoid arthritis. VIGOR Study Group. N Engl J Med. 2000 Nov 23;343(21):1520-8, 2 p following 1528. doi: 10.1056/NEJM200011233432103. PMID 11087881
- [Background] Colombel M, Saint F, Chopin D, Malavaud B, Nicolas L, Rischmann P. The effect of ofloxacin on bacillus calmette-guerin induced toxicity in patients with superficial bladder cancer: results of a randomized, prospective, double-blind, placebo controlled, multicenter study. J Urol. 2006 Sep;176(3):935-9. doi: 10.1016/j.juro.2006.04.104. PMID 16890660
- [Background] Dovedi SJ, Kirby JA, Davies BR, Leung H, Kelly JD. Celecoxib has potent antitumour effects as a single agent and in combination with BCG immunotherapy in a model of urothelial cell carcinoma. Eur Urol. 2008 Sep;54(3):621-30. doi: 10.1016/j.eururo.2008.01.013. Epub 2008 Jan 15. PMID 18222600
- [Background] Grubbs CJ, Lubet RA, Koki AT, Leahy KM, Masferrer JL, Steele VE, Kelloff GJ, Hill DL, Seibert K. Celecoxib inhibits N-butyl-N-(4-hydroxybutyl)-nitrosamine-induced urinary bladder cancers in male B6D2F1 mice and female Fischer-344 rats. Cancer Res. 2000 Oct 15;60(20):5599-602. PMID 11059745
- [Background] Kilbridge KL, Kantoff P. Intravesical therapy for superficial bladder cancer: is it a wash? J Clin Oncol. 1994 Jan;12(1):1-4. doi: 10.1200/JCO.1994.12.1.1. No abstract available. PMID 8270966
- [Background] Klein RD, Van Pelt CS, Sabichi AL, Dela Cerda J, Fischer SM, Furstenberger G, Muller-Decker K. Transitional cell hyperplasia and carcinomas in urinary bladders of transgenic mice with keratin 5 promoter-driven cyclooxygenase-2 overexpression. Cancer Res. 2005 Mar 1;65(5):1808-13. doi: 10.1158/0008-5472.CAN-04-3567. PMID 15753378
- [Background] Koya MP, Simon MA, Soloway MS. Complications of intravesical therapy for urothelial cancer of the bladder. J Urol. 2006 Jun;175(6):2004-10. doi: 10.1016/S0022-5347(06)00264-3. PMID 16697786
- [Background] Malmstrom PU, Wijkstrom H, Lundholm C, Wester K, Busch C, Norlen BJ. 5-year followup of a randomized prospective study comparing mitomycin C and bacillus Calmette-Guerin in patients with superficial bladder carcinoma. Swedish-Norwegian Bladder Cancer Study Group. J Urol. 1999 Apr;161(4):1124-7. PMID 10081852
- [Background] Miyata Y, Kanda S, Nomata K, Eguchi J, Kanetake H. Expression of cyclooxygenase-2 and EP4 receptor in transitional cell carcinoma of the upper urinary tract. J Urol. 2005 Jan;173(1):56-60. doi: 10.1097/01.ju.0000148272.77539.2d. PMID 15592025
- [Background] Phillips RK, Wallace MH, Lynch PM, Hawk E, Gordon GB, Saunders BP, Wakabayashi N, Shen Y, Zimmerman S, Godio L, Rodrigues-Bigas M, Su LK, Sherman J, Kelloff G, Levin B, Steinbach G; FAP Study Group. A randomised, double blind, placebo controlled study of celecoxib, a selective cyclooxygenase 2 inhibitor, on duodenal polyposis in familial adenomatous polyposis. Gut. 2002 Jun;50(6):857-60. doi: 10.1136/gut.50.6.857. PMID 12010890
- [Background] Ristimaki A, Nieminen O, Saukkonen K, Hotakainen K, Nordling S, Haglund C. Expression of cyclooxygenase-2 in human transitional cell carcinoma of the urinary bladder. Am J Pathol. 2001 Mar;158(3):849-53. doi: 10.1016/S0002-9440(10)64033-3. PMID 11238034
- [Background] Serretta V, Pavone C, Ingargiola GB, Daricello G, Allegro R, Pavone-Macaluso M. TUR and adjuvant intravesical chemotherapy in T1G3 bladder tumors: recurrence, progression and survival in 137 selected patients followed up to 20 years. Eur Urol. 2004 Jun;45(6):730-5; discussion 735-6. doi: 10.1016/j.eururo.2003.12.002. PMID 15149744
- [Background] Shariat SF, Kim JH, Ayala GE, Kho K, Wheeler TM, Lerner SP. Cyclooxygenase-2 is highly expressed in carcinoma in situ and T1 transitional cell carcinoma of the bladder. J Urol. 2003 Mar;169(3):938-42. doi: 10.1097/01.ju.0000043638.89552.ed. PMID 12576817
- [Background] Shelley MD, Kynaston H, Court J, Wilt TJ, Coles B, Burgon K, Mason MD. A systematic review of intravesical bacillus Calmette-Guerin plus transurethral resection vs transurethral resection alone in Ta and T1 bladder cancer. BJU Int. 2001 Aug;88(3):209-16. doi: 10.1046/j.1464-410x.2001.02306.x. PMID 11488731
- [Background] Solomon SD, McMurray JJ, Pfeffer MA, Wittes J, Fowler R, Finn P, Anderson WF, Zauber A, Hawk E, Bertagnolli M; Adenoma Prevention with Celecoxib (APC) Study Investigators. Cardiovascular risk associated with celecoxib in a clinical trial for colorectal adenoma prevention. N Engl J Med. 2005 Mar 17;352(11):1071-80. doi: 10.1056/NEJMoa050405. Epub 2005 Feb 15. PMID 15713944
- [Background] Steinbach G, Lynch PM, Phillips RK, Wallace MH, Hawk E, Gordon GB, Wakabayashi N, Saunders B, Shen Y, Fujimura T, Su LK, Levin B, Godio L, Patterson S, Rodriguez-Bigas MA, Jester SL, King KL, Schumacher M, Abbruzzese J, DuBois RN, Hittelman WN, Zimmerman S, Sherman JW, Kelloff G. The effect of celecoxib, a cyclooxygenase-2 inhibitor, in familial adenomatous polyposis. N Engl J Med. 2000 Jun 29;342(26):1946-52. doi: 10.1056/NEJM200006293422603. PMID 10874062
- [Background] Sylvester RJ, van der Meijden AP, Oosterlinck W, Witjes JA, Bouffioux C, Denis L, Newling DW, Kurth K. Predicting recurrence and progression in individual patients with stage Ta T1 bladder cancer using EORTC risk tables: a combined analysis of 2596 patients from seven EORTC trials. Eur Urol. 2006 Mar;49(3):466-5; discussion 475-7. doi: 10.1016/j.eururo.2005.12.031. Epub 2006 Jan 17. PMID 16442208
- [Background] Sylvester RJ, Oosterlinck W, Witjes JA. The schedule and duration of intravesical chemotherapy in patients with non-muscle-invasive bladder cancer: a systematic review of the published results of randomized clinical trials. Eur Urol. 2008 Apr;53(4):709-19. doi: 10.1016/j.eururo.2008.01.015. Epub 2008 Jan 15. PMID 18207317
- [Background] van Rhijn BW, Burger M, Lotan Y, Solsona E, Stief CG, Sylvester RJ, Witjes JA, Zlotta AR. Recurrence and progression of disease in non-muscle-invasive bladder cancer: from epidemiology to treatment strategy. Eur Urol. 2009 Sep;56(3):430-42. doi: 10.1016/j.eururo.2009.06.028. Epub 2009 Jun 26. PMID 19576682
- [Background] Witjes JA, Hendricksen K. Intravesical pharmacotherapy for non-muscle-invasive bladder cancer: a critical analysis of currently available drugs, treatment schedules, and long-term results. Eur Urol. 2008 Jan;53(1):45-52. doi: 10.1016/j.eururo.2007.08.015. Epub 2007 Aug 20. PMID 17719169